CLINICAL TRIAL: NCT02454998
Title: The Difference in the Surgical Outcome of Unilateral Cleft Lip and Palate Between Patients With and Without Pre-Alveolar Bone Graft Orthodontic Treatment
Brief Title: Alveolar Bone Grafting Outcome Between Patient With and Without Orthodontic Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 102-3500C (99-3910A3); CMRPG3B0201-3 (Other Grant/Funding Number: Chang Gung Memorial Hospital research grant)
Record Dates: First submitted 2015-02-17; First posted 2015-05-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-02

CONDITIONS: Cleft Lip
Keywords: Unilateral complete cleft lip; Alveolar bone graft
MeSH Terms: conditions — Cleft Lip | interventions — Orthodontics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Orthodontic treatment arm (Experimental): Previous to the surgical alveolar bone grafting, orthodontic treatment is performed several months before surgery
  Interventions: Other: orthodontic treatment
- No orthodontic treatment arm (No Intervention): No orthodontic treatment previous to surgical alveolar bone grafting

INTERVENTIONS:
Other: orthodontic treatment — Braces on the upper dental arch previous to surgical alveolar bone grafting. the goal is optimizing the structure of dental-alveolar structure.
  Arms: Orthodontic treatment arm

SUMMARY:
Alveolar bone grafting (ABG) is an essential part of the surgical management of cleft lip and palate patients. This procedure could obliterate oronasal fistula, stabilize dental arch, offer bone matrix for adjacent teeth eruption. Moreover, by obliterating oronasal fistula, we stop the chronic irritation of nasal mucosa by oral content. Hence, the symptoms of rhinorrhea or nasal obstruction could be improved. This dental arch defect could predispose further dental arch medial collapse. Without alveolar bone grafting the dental arch is not stable, dental movement during orthodontic treatment is limited and dental arch expansion is not possible.

Previous to operation, the patient suffered from dental crowding and dental inclination toward to the cleft. This produces a difficult dental hygiene and predispose to dental caries and gingivitis. Pre-operative orthodontics treatment is advised in many centers. By aligned the teeth previous to surgery, with a better dental hygiene, we purpose that the infection rate will be reduced and success rate will be better.

The Purpose of this study is to determine whether pre-operative orthopedic treatment will affect secondary alveolar bone grafting outcome and to assess the nasal change after alveolar bone graft.

DETAILED DESCRIPTION:
Overall goals of study:

The goals of this study are to determine whether pre-operative orthodontic treatment will affect secondary alveolar bone grafting outcome

Importance of alveolar bone grafting Alveolar bone cleft is present in the majority of patients with cleft lip and palate. This bone cleft destabilizes the maxillary arch and predisposes it to medial collapse. Teeth will not erupt in this region of alveolar bone defect. Permanent stabilization of the maxillary segments into a functional dental arch form is achieved by reconstruction of alveolar with bone grafts. The goals of alveolar bone grafting are to maintain normal occlusion and to provide a matrix for the continued eruption of permanent teeth in this region. Moreover, future maxillary expansion cannot be done unless repair of the alveolar cleft is coordinated with the desired orthodontic movement.

Timing of alveolar bone grafting Maxillary growth and dental age are the predominant considerations in determining the timing of alveolar reconstruction. Maxillary growth is completed near the age of eight years old, whereas the maxillary canine does not erupt before the age of ten.Therefore, to minimize growth disturbance to the maxilla, reconstruction should be performed after the growth is completed.It has been widely agreed that the timing of alveolar grafting should be around the stage of mixed dentition . The bone grafting should be completed at approximately nine years of age when the bulk of the alveolar bone growth is completed and the incisors are erupted, while the lateral incisors and canines are starting to erupt into alveolar cleft region

Diagnosis Radiographic studies, including panoramic radiographs, selected periapical films, Cephalographic films and recently CT scan are integral parts for diagnosis and evaluation. They provide important assessments of the pre-operative dentition in the vicinity of the cleft, the dimensions and structures of cleft itself as well as postoperative condition of the bone bridge after alveolar bone grafting.The CT scan offers more detailed pre-operative and post-operative bone structures with less distortion. Additionally, CT scan also provide: 1. Detailed information about the depth and volume of bone deposited in the cleft, 2. More consistent in showing bone trabeculation, 3. Detailed position of erupting teeth relative to the bone graft, 4. More detailed bone and teeth anatomy for clinical orthodontics decisions. In addition, the CT scan could offer 3D lineal measurements and volumetric analysis . Arai et al. developed a novel cone-bean CT (CBCT) or Ortho CT which has important characteristics such as lowered radiation dose and the ability to produce higher resolution compared to conventional spiral CT. Several reports have indicated that it is clinical useful for the 3D imaging diagnosis in the maxillofacial region.

Pre-operative orthodontic treatment The orthodontists form an integral part in the cleft care. Their recommendations regarding timing of treatment should be carefully considered before surgical treatment. The dental crowding and malposition of the teeth around the cleft can interfere with oral hygiene . The goal of the preoperative orthodontic treatment is to optimizing the position of dentoalveolar structure which enables the patients to have better oral hygiene prior to the operation. Some centers have recommended that the orthodontic treatment become part of the treatment protocol for their patients However, the presurgical orthodontics treatment is time consuming as the children are required to visit the clinic for monthly orthodontic adjustment. The average duration of the orthodontic treatments before operation is 6 months. These factors not only add discomfort to the children but also create significant financial burden to the parents. Even this primary orthodontic treatment is able to align the upper dental arch; secondary orthodontic treatment is always needed after complete permanent teeth eruption. Therefore, the actual need of presurgical orthodontics remained questionable. No studies have yet to actually address the outcome of alveolar bone grafting with or without presurgical orthodontics. The primary goal of this present prospective randomize study is to determine whether pre-operative orthodontics treatment will affect secondary alveolar bone grafting outcome.

Donor site selection:

The bones used most commonly include the iliac crest, calvarial or tibia. Regardless of the donor site, cancellous bone is preferable to cortical or osteochondral graft . The iliac crest as a donor site is preferred because it has sufficient cancellous bone to fill even a large alveolar bone defect.

Surgical procedures:

The surgical procedures of alveolar bone graft are similar to the procedures that were described by Hall and Posnick et al. except with some minor modifications. With adequate general anesthesia via orotracheal intubation, two teams worked at the same time with one team harvesting the bone graft and the other team preparing the recipient site at the oral cavity. Attention was turned to the right hip where an oblique incision was made lateral and parallel to the iliac crest. The incision was deepened to the periosteum of the lateral cortex. The iliac crest was reflected medially as a bone flap. Cancellous bone chips was harvested. At the same time, the other team was working on the oral cavity. The mouth was suctioned and a throat pack was placed. The gingiva and upper buccal sulcus were infiltrated with 1% Xylocaine in 1:200,000 epinephrine solutions for hemostasis and easier dissection. Incisions were made along each side of the alveolar cleft. A superiorly based gingival mucoperiosteal flap was designed and raised sharply from the gingival margin on the lesser segment. The flap was extended posteriorly to the first molar. The incision was then curved up obliquely towards the buccal sulcus. The flap on the medial segment was elevated in a similar fashion towards the midline. The palatal mucoperiosteal flaps were raised to a level beyond the deepest margin of the alveolar fistula. The fistula margins at the palatal side were freshened and sutured. The nasal floor tissue could be completely separated from the palatal mucoperiosteum after raising the palatal flaps and could then be stripped off the bony cleft. The nasal floor tissue was dissected upward reaching the pyriform aperture on the lateral segment and the cartilaginous septum on the medial segment. This allowed a tension-free closure of nasal floor tissue and adequate correction of the vertical discrepancy of the nostril sill. The nasal floor fistula was securely repaired with 4-0 Vicryl sutures. Cancellous bone chips which were already harvested from iliac bone by another team were packed firmly into the bony defect to the level of the alveolar process and the pyriform aperture on the cleft side. The periosteum of the lateral gingival flap was scored to reduce the tension especially at the lateral end of the incision. The lateral gingival flap was then advanced and sutured to the medial flap and palatal flap to provide a watertight and tension free closure.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral complete cleft lip patients
2. Alveolar bone cleft diagnosed with conventional radiographic study
3. Patients at the stage of mixed dentition.
4. Informed consent signed by the parents or custodians.

Exclusion Criteria:

1. Presentation of other craniofacial anomalies.
2. Parents or custodians who do not agreed to this procedure.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2011-02; Primary Completion 2015-07 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Pre-orthodontic alveolar bone defect | Before surgical and orthodontic treatment, A expected average of 6 months before surgery
  CT scan, measurement of alveolar bone cleft defect volume
Pre-surgical alveolar bone defect | Before surgical treatment (alveolar bone cleft), a expected average of 6 months of orthodontic treatment
  CT scan, measurement of alveolar bone cleft defect volume
Alveolar bone graft survival | A expected average of 6 months after surgery
  CT scan, measurement of volume of bone graft filling the alveolar bone cleft

SECONDARY OUTCOMES:
Infection rate | up to 6 months
  Evaluate the infection rate after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Philip Kuo-Ting Chen, M.D., Study Chair — Chang Gung Memorial Hospital

REFERENCES:
- [Background] Abyholm FE, Bergland O, Semb G. Secondary bone grafting of alveolar clefts. A surgical/orthodontic treatment enabling a non-prosthodontic rehabilitation in cleft lip and palate patients. Scand J Plast Reconstr Surg. 1981;15(2):127-40. doi: 10.3109/02844318109103425. No abstract available. PMID 7041248
- [Background] Boyne PJ, Sands NR. Secondary bone grafting of residual alveolar and palatal clefts. J Oral Surg. 1972 Feb;30(2):87-92. No abstract available. PMID 4550446
- [Background] Bajaj AK, Wongworawat AA, Punjabi A. Management of alveolar clefts. J Craniofac Surg. 2003 Nov;14(6):840-6. doi: 10.1097/00001665-200311000-00005. PMID 14600625
- [Background] da Silva Filho OG, Boiani E, de Oliveira Cavassan A, Santamaria M Jr. Rapid maxillary expansion after secondary alveolar bone grafting in patients with alveolar cleft. Cleft Palate Craniofac J. 2009 May;46(3):331-8. doi: 10.1597/07-205.1. Epub 2008 Oct 29. PMID 19642749
- [Background] Sato Y, Grayson BH, Garfinkle JS, Barillas I, Maki K, Cutting CB. Success rate of gingivoperiosteoplasty with and without secondary bone grafts compared with secondary alveolar bone grafts alone. Plast Reconstr Surg. 2008 Apr;121(4):1356-1367. doi: 10.1097/01.prs.0000302461.56820.c9. PMID 18349656
- [Background] Hsieh CH, Ko EW, Chen PK, Huang CS. The effect of gingivoperiosteoplasty on facial growth in patients with complete unilateral cleft lip and palate. Cleft Palate Craniofac J. 2010 Sep;47(5):439-46. doi: 10.1597/08-207. PMID 20180706
- [Background] Witherow H, Cox S, Jones E, Carr R, Waterhouse N. A new scale to assess radiographic success of secondary alveolar bone grafts. Cleft Palate Craniofac J. 2002 May;39(3):255-60. doi: 10.1597/1545-1569_2002_039_0255_anstar_2.0.co_2. PMID 12019000
- [Background] Bergland O, Semb G, Abyholm FE. Elimination of the residual alveolar cleft by secondary bone grafting and subsequent orthodontic treatment. Cleft Palate J. 1986 Jul;23(3):175-205. PMID 3524905
- [Background] Jia YL, Fu MK, Ma L. Long-term outcome of secondary alveolar bone grafting in patients with various types of cleft. Br J Oral Maxillofac Surg. 2006 Aug;44(4):308-12. doi: 10.1016/j.bjoms.2005.07.003. Epub 2005 Aug 16. PMID 16107298
- [Background] Craven C, Cole P, Hollier L Jr, Stal S. Ensuring success in alveolar bone grafting: a three-dimensional approach. J Craniofac Surg. 2007 Jul;18(4):855-9. doi: 10.1097/scs.0b013e31806849fa. PMID 17667677
- [Background] Enemark H, Sindet-Pedersen S, Bundgaard M. Long-term results after secondary bone grafting of alveolar clefts. J Oral Maxillofac Surg. 1987 Nov;45(11):913-9. doi: 10.1016/0278-2391(87)90439-3. PMID 3312537
- [Background] Sindet-Pedersen S, Enemark H. Comparative study of secondary and late secondary bone-grafting in patients with residual cleft defects. Short-term evaluation. Int J Oral Surg. 1985 Oct;14(5):389-98. doi: 10.1016/s0300-9785(85)80071-5. PMID 3932232
- [Background] Honma K, Kobayashi T, Nakajima T, Hayasi T. Computed tomographic evaluation of bone formation after secondary bone grafting of alveolar clefts. J Oral Maxillofac Surg. 1999 Oct;57(10):1209-13. doi: 10.1016/s0278-2391(99)90488-3. PMID 10513867
- [Background] Tai CC, Sutherland IS, McFadden L. Prospective analysis of secondary alveolar bone grafting using computed tomography. J Oral Maxillofac Surg. 2000 Nov;58(11):1241-9; discussion 1250. doi: 10.1053/joms.2000.16623. PMID 11078135
- [Background] Hamada Y, Kondoh T, Noguchi K, Iino M, Isono H, Ishii H, Mishima A, Kobayashi K, Seto K. Application of limited cone beam computed tomography to clinical assessment of alveolar bone grafting: a preliminary report. Cleft Palate Craniofac J. 2005 Mar;42(2):128-37. doi: 10.1597/03-035.1. PMID 15748103
- [Background] Waitzman AA, Posnick JC, Armstrong DC, Pron GE. Craniofacial skeletal measurements based on computed tomography: Part I. Accuracy and reproducibility. Cleft Palate Craniofac J. 1992 Mar;29(2):112-7. doi: 10.1597/1545-1569_1992_029_0112_csmboc_2.3.co_2. PMID 1571344
- [Background] Goudy S, Lott D, Burton R, Wheeler J, Canady J. Secondary alveolar bone grafting: outcomes, revisions, and new applications. Cleft Palate Craniofac J. 2009 Nov;46(6):610-2. doi: 10.1597/08-126.1. Epub 2009 May 19. PMID 19860505